CLINICAL TRIAL: NCT06421532
Title: A Partial Randomised Clinical Trial Investigating Stimulation of the Glymphatic System by Either Deepening Sleep With Lower-sodium Oxybate or Inhibiting Cortical Spreading Depressions With Non-invasive Vagus Nerve Stimulation, or Both, in Patients With Cerebral Amyloid Angiopathy (CAA)
Brief Title: Stimulating Amyloid Clearance in Cerebral Amyloid Angiopathy
Acronym: Clear-Brain
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: The Dutch Brain Foundation (Other)
Responsible Party: Principal Investigator, Rolf Fronczek, principal investigator and neurologist, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P23.100
Record Dates: First submitted 2024-05-08; First posted 2024-05-20 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-08

CONDITIONS: Cerebral Amyloid Angiopathy
MeSH Terms: conditions — Cerebral Amyloid Angiopathy

STUDY DESIGN:
Intervention Model Description: pre-post study with additional randomisation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Low-sodium oxybate (LXB) (Experimental): Deepening sleep
  Interventions: Drug: XYWAV
- Non-invasive vagus nerve stimulation (nVNS) (Experimental): Inhibiting cortical spreading depolarisations
  Interventions: Device: gammaCore Sapphire
- Combination of both (Experimental): Deepening sleep and inhibiting cortical spreading depolarisations
  Interventions: Drug: XYWAV; Device: gammaCore Sapphire

INTERVENTIONS:
Drug: XYWAV — Daily before bedtime for 3 months
  Arms: Combination of both; Low-sodium oxybate (LXB)
Device: gammaCore Sapphire — Twice daily for 3 months
  Arms: Combination of both; Non-invasive vagus nerve stimulation (nVNS)

SUMMARY:
A pre-post study will be conducted to assess whether treatment with LXB, nVNS or a combination of both interventions can enhance the clearance of Aβ in patients with CAA. A total of 60 subjects, 30 with sCAA and 30 with D-CAA, will be randomly assigned to receive LXB, or both interventions. The primary outcome measure will be the morning levels of Aβ40 and Aβ42 in cerebrospinal fluid (CSF) before and after the intervention. The investigators will assess disease progression with (non-)haemorrhagic imaging markers on 7-Tesla Magnetic Resonance Imaging (7-T MRI) as a secondary outcome. Additionally, the activity of the glymphatic system by means of fluid dynamics will be assessed using 7-T MRI.

ELIGIBILITY:
Inclusion Criteria:

* Patients with D-CAA with a proven amyloid precursor protein (APP) mutation or a history of ≥1 lobar intracerebral haemorrhage (ICH) and a positive family history for D-CAA in ≥1 first degree relative

  * Age ≥30 years old
  * ≤ 2 symptomatic ICH (occurrence of ICH at least > 1 year ago) or presence of ≥ 1 haemorrhagic marker (cortical superficial siderosis, cerebral microbleeds) or non-haemorrhagic marker (white matter hyperintensities, enlarged perivascular spaces).
  * When presymptomatic, patients are aware that they have D-CAA
* Probable sporadic CAA (sCAA) according to the Modified Boston criteria 2.0

  * Age ≥50 years old
  * ≤ 2 symptomatic ICH (occurrence of ICH at least > 1 year ago)
* Provisional CAA when the criteria for probable sCAA are not met due to presence of deep haemorrhagic lesions but there are mostly lobar microbleeds (MBs) and cortical superficial siderosis (cSS) present or a ratio of 10 times more lobar MBs than deep MBs without cSS.

  * Age ≥50 years old
  * ≤ 2 symptomatic ICH (occurrence of ICH at least > 1 year ago)
* Participants able to read and understand the patient information folder and who freely provide written informed consent

Exclusion Criteria:

* Modified Rankin Score ≥ 4
* A life expectancy of less than six months
* Pregnancy/breast feeding
* Contraindications for lumbar puncture
* Unwillingness to refrain from consuming > 1 alcohol unit per day and not later than 8 pm, during the intervention period.

Contraindications for using LXB:

* Sleep apnea; patients will be screened with respiratory polygraphy before inclusion and screening by questionnaire during intervention with LXB.
* Restless legs (RLS) needing active treatment with RLS medication.
* Currently suffering from severe depression and using medication or receiving cognitive therapy.
* Porphyria
* Succinic semialdehyde dehydrogenase (SSADH-)deficiency
* Use of opiates, barbiturates, sedatives (dexmedetomidine, temazepam, oxazepam, midazolam)
* Use certain medication before inclusion:

  * When benzodiazepine is used: a two nights washout before the intervention (T3) will be started, is needed.
  * When LXB or SXB is used before inclusion: one week washout before inclusion and no use of LXB or SXB during inclusion except for the intervention dose.

Contraindications for lumbar puncture:

* Compression of the spinal cord
* Signs and symptoms of increased intracranial pressure
* Local infections of the skin at the puncture site
* Coagulopathy or thrombocytopenia (<100)
* (Use of acetylsalicylic acid, NSAIDs, COX2 inhibitors or prophylactic low-molecular-weight heparin are no contraindications for lumbar puncture.)
* Participants deemed at risk for brain replacement due to known aqueduct stenosis, Arnold chiari malformations.
* Participants with a lumbo-sacral neural tube defect or who have a ventriculo-atrial or ventriculo-peritoneal drain.

Contraindications for nVNS:

* An active implantable medical device such as a pacemaker, deep brain stimulator, or any implanted electronic device.
* A recent (< 1 month) brain infarction or transient ischemic attack due to a symptomatic stenosis or dissection of the carotid artery (in these patients the other side will be stimulated unless a significant stenosis or dissection on the other side is present as well).
* If someone knows to have a structural abnormality e.g. lymphadenopathy, previous surgery or abnormal anatomy (in these patients the other side will be stimulated)
* Metal cervical spine hardware or metallic implant near the stimulation site
* Cervical vagotomy (in these patients the other side will be stimulated)

Contraindications for 7 Tesla MRI as determined by the 7 Tesla safety committee. Examples of possible contra-indications are:

* Claustrophobia
* Pacemakers and defibrillators
* Nerve stimulators
* Intracranial clips
* Intraorbital or intraocular metallic fragments
* Cochlear implants
* Ferromagnetic implants
* Hydrocephalus pump
* Intra-uterine device
* Permanent make-up
* Tattoos above the shoulders

Specific contraindications for checkerboard functional Magnetic Resonance Imaging (fMRI):

* Seizure within prior year
* Photosensitive epilepsy
* Non-correctable visual impairment

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-27 (Actual); Primary Completion 2027-09-27 (Estimated); Study Completion 2027-09-27 (Estimated)

PRIMARY OUTCOMES:
Amyloid-beta 40 and 42 in cerebrospinal fluid | 3 months
  Difference between before and after intervention

SECONDARY OUTCOMES:
Disease progression with (non-)haemorrhagic imaging markers on 7-T MRI | 2x 3 months
  Intracerebral haemorrhages, cerebral microbleeds, cortical superficial siderosis, white matter hyperintensities, perivascular spaces, cerebrovascular reactivity
Other liquid biomarkers | 3 months
  Levels of amyloid-beta 38, 43, t-tau and p-tau181 in CSF and levels of amyloid-beta 40 and 42 in serum.
Activity of the glymphatic system by means of fluid dynamics on 7-T MRI | 2x 3 months
  CSF motion

CONTACTS AND LOCATIONS:
Locations (1):
- Leiden University Medical Center (LUMC), Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No